CLINICAL TRIAL: NCT03670186
Title: Effects of BDNF Val66Met Polymorphism on the Efficacy of Aerobic Exercise in Sedentary, Healthy Males
Brief Title: Effects of Genetic Variation on the Efficacy of Aerobic Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: BDNF V66M Exercise Study
Record Dates: First submitted 2018-09-05; First posted 2018-09-13 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Quality of Life
MeSH Terms: interventions — High-Intensity Interval Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- V66V-HIIT (Experimental): Val/Val carriers who undergo high-intensity interval training (HIIT) for 6 weeks, 3 times per week
  Interventions: Behavioral: High-Intensity Interval Training (HIIT)
- V66M-HIIT (Experimental): Val/Met carriers who undergo high-intensity interval training (HIIT) for 6 weeks, 3 times per week
  Interventions: Behavioral: High-Intensity Interval Training (HIIT)

INTERVENTIONS:
Behavioral: High-Intensity Interval Training (HIIT) — Participants perform high-intensity interval training (HIIT) on a cycle ergometer. The HIIT protocol consists of a 3-minute warm-up at 50W, ten 60-second high-intensity cycling intervals interspersed with 90 seconds of active recovery at 30% of their peak power output and a 2-minute cool-down at 50W for a total of 17.5 minutes.

SUMMARY:
This study investigates whether, after six weeks of exercise, a genetic variant (Val66Met) in the gene that makes a molecule (BDNF) important for brain health and function, influences the beneficial effects of a further session of exercise in sedentary, healthy males. The aim of this research is to determine whether not having this genetic variant (Val66Met) provides an advantage for achieving greater exercise-induced benefits. After six consecutive weeks of exercise (high-intensity interval training (HIIT), three times per week), the effects of a further session of exercise on brain activity are studied in healthy, sedentary males with and without the BDNF genetic variant. Further, whether the BDNF genetic variant impacts the effects of six weeks of aerobic exercise on blood BDNF levels, memory and cardiorespiratory fitness is examined. This data will help to understand whether genetic factors moderate the beneficial effects of exercise. Understanding what factors influence the effectiveness of exercise training programs is essential to individualize exercise programs and maximize their positive effects on the brain and during rehabilitation following brain injuries.

DETAILED DESCRIPTION:
Aerobic exercise promotes brain health and function. Indeed, exercise has been shown to improve learning and memory, delay cognitive decline and protect against brain atrophy in healthy aging individuals. Additionally, exercise programs reduce brain injury and delay onset and progression of neurodegenerative diseases such as Alzheimer's. However, individual variability in the efficacy of these programs limit their widespread application as a "therapeutic". Genetic variants may contribute to the large degree of individual variability in the effects of exercise on cognition and brain health.

Brain-derived neurotrophic factor (BDNF) is a neurotrophin that plays a key role in activity-dependent neuroplasticity. Rodent studies show that increases in BDNF mediate the effects of exercise on learning and memory. A single nucleotide polymorphism in the BDNF gene that causes a valine (Val) to methionine (Met) substitution at codon 66 reduces activity-dependent secretion of BDNF and is associated with altered hippocampal activation and poorer episodic memory. The objective of this research is to determine whether after six consecutive weeks of high-intensity interval training (HIIT), three times per week, BDNF Val66Met polymorphism impacts the effects of a further HIIT session on corticospinal excitability as well as intracortical and spinal circuitry. Additionally, this study aims to assess whether BDNF Val66Met polymorphism moderates the effects of six consecutive weeks of HIIT on BDNF, working memory and cardiorespiratory fitness levels. The findings will indicate whether the BDNF Val allele provides an advantage for achieving greater exercise-induced benefits and could thus help individualize exercise programs to maximize their beneficial effects. These data will also provide insights into the mechanisms by which aerobic exercise induces neuroplasticity.

ELIGIBILITY:
Inclusion Criteria:

1. do not engage or engage in less than or equal to 60 minutes of structured exercise per week (or two exercise sessions of 30 min/week; Heisz et al., 2017; Little et al. 2011) as per their self-report;
2. must be able to engage in physical activity and thus must answer 'NO' to all questions on the Get Active Questionnaire (GAQ). If potential participants answer 'YES' to any of the GAQ questions, they are immediately deemed ineligible to partake in the research;
3. must not take street drugs and medications, including alpha blockers, antibiotics, antipsychotics, benzodiazepines, beta-blockers, calcium channel blockers, systemic corticosteroids, muscle relaxants, neuromuscular blocking agents, sedatives, and psychostimulants, and must have no stable or unstable medical conditions, history of neurological or psychological disorders, head injury and/or surgery, seizures or have a family history of seizures or epilepsy, experience frequent headaches, migraines and sleep deprivation as per the TMS screening form;
4. must be right-handed as per the handedness questionnaire;
5. must be between 18 and 30 years old.

Exclusion Criteria:

1. engage in more than 60 minutes of structured exercise per week (or two exercise sessions of 30 min/week; Heisz et al., 2017; Little et al. 2011) as per their self-report;
2. are not able to engage in physical activity and thus answer 'YES' to any of the GAQ questions;
3. take street drugs and medications, including alpha blockers, antibiotics, antipsychotics, benzodiazepines, beta-blockers, calcium channel blockers, systemic corticosteroids, muscle relaxants, neuromuscular blocking agents, sedatives, and psychostimulants, and must have no stable or unstable medical conditions, history of neurological or psychological disorders, head injury and/or surgery, seizures or have a family history of seizures or epilepsy, experience frequent headaches, migraines and sleep deprivation as per the TMS screening form;
4. are not right-handed as per the handedness questionnaire;
5. are younger than 18 years of age and older than 30 years of age.

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2018-12-03 (Actual); Study Completion 2019-01-21 (Actual)

PRIMARY OUTCOMES:
Corticospinal excitability | 8 weeks
  Corticospinal excitability as measured by single-pulse TMS-evoked responses in a hand and forearm muscles.
Intracortical circuits | 8 weeks
  Intracortical circuits as measured by paired-pulse TMS-evoked responses in a hand muscle
Spinal circuits | 8 weeks
  Spinal circuits as measured by spinal Hoffman reflexes from a forearm muscle
Blood BDNF | 8 weeks
  Serum levels of BDNF as assessed by ELISA

SECONDARY OUTCOMES:
Cathepsin B | 8 weeks
  Serum levels of cathepsin B as assessed by ELISA
IGF-1 | 8 weeks
  Serum levels of IGF-1 as assessed by ELISA
VEGF | 8 weeks
  Serum levels of VEGF as assessed by ELISA
Osteocalcin | 8 weeks
  Serum levels of osteocalcin as assessed by ELISA
Working memory | 8 weeks
  Working memory as assessed by the Automated Operation Span (OSPAN) Task
Cardiorespiratory fitness | 8 weeks
  Cardiorespiratory fitness as assessed by VO2 peak test

CONTACTS AND LOCATIONS:
Overall Officials: Aimee Nelson, PhD, Principal Investigator — McMaster University
Locations (1):
- McMaster University, Ivor Wynne Centre (IWC) building, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Begliuomini S, Casarosa E, Pluchino N, Lenzi E, Centofanti M, Freschi L, Pieri M, Genazzani AD, Luisi S, Genazzani AR. Influence of endogenous and exogenous sex hormones on plasma brain-derived neurotrophic factor. Hum Reprod. 2007 Apr;22(4):995-1002. doi: 10.1093/humrep/del479. Epub 2007 Jan 24. PMID 17251358
- [Background] Colcombe S, Kramer AF. Fitness effects on the cognitive function of older adults: a meta-analytic study. Psychol Sci. 2003 Mar;14(2):125-30. doi: 10.1111/1467-9280.t01-1-01430. PMID 12661673
- [Background] Egan MF, Kojima M, Callicott JH, Goldberg TE, Kolachana BS, Bertolino A, Zaitsev E, Gold B, Goldman D, Dean M, Lu B, Weinberger DR. The BDNF val66met polymorphism affects activity-dependent secretion of BDNF and human memory and hippocampal function. Cell. 2003 Jan 24;112(2):257-69. doi: 10.1016/s0092-8674(03)00035-7. PMID 12553913
- [Background] Heisz JJ, Clark IB, Bonin K, Paolucci EM, Michalski B, Becker S, Fahnestock M. The Effects of Physical Exercise and Cognitive Training on Memory and Neurotrophic Factors. J Cogn Neurosci. 2017 Nov;29(11):1895-1907. doi: 10.1162/jocn_a_01164. Epub 2017 Jul 12. PMID 28699808
- [Background] Itoh K, Hashimoto K, Kumakiri C, Shimizu E, Iyo M. Association between brain-derived neurotrophic factor 196 G/A polymorphism and personality traits in healthy subjects. Am J Med Genet B Neuropsychiatr Genet. 2004 Jan 1;124B(1):61-3. doi: 10.1002/ajmg.b.20078. PMID 14681916
- [Background] Lamy JC, Russmann H, Shamim EA, Meunier S, Hallett M. Paired associative stimulation induces change in presynaptic inhibition of Ia terminals in wrist flexors in humans. J Neurophysiol. 2010 Aug;104(2):755-64. doi: 10.1152/jn.00761.2009. Epub 2010 Jun 10. PMID 20538768
- [Background] Little JP, Gillen JB, Percival ME, Safdar A, Tarnopolsky MA, Punthakee Z, Jung ME, Gibala MJ. Low-volume high-intensity interval training reduces hyperglycemia and increases muscle mitochondrial capacity in patients with type 2 diabetes. J Appl Physiol (1985). 2011 Dec;111(6):1554-60. doi: 10.1152/japplphysiol.00921.2011. Epub 2011 Aug 25. PMID 21868679
- [Background] Lommatzsch M, Zingler D, Schuhbaeck K, Schloetcke K, Zingler C, Schuff-Werner P, Virchow JC. The impact of age, weight and gender on BDNF levels in human platelets and plasma. Neurobiol Aging. 2005 Jan;26(1):115-23. doi: 10.1016/j.neurobiolaging.2004.03.002. PMID 15585351
- [Background] Lu B, Chow A. Neurotrophins and hippocampal synaptic transmission and plasticity. J Neurosci Res. 1999 Oct 1;58(1):76-87. PMID 10491573
- [Background] Lulic T, El-Sayes J, Fassett HJ, Nelson AJ. Physical activity levels determine exercise-induced changes in brain excitability. PLoS One. 2017 Mar 9;12(3):e0173672. doi: 10.1371/journal.pone.0173672. eCollection 2017. PMID 28278300
- [Background] Neeper SA, Gomez-Pinilla F, Choi J, Cotman C. Exercise and brain neurotrophins. Nature. 1995 Jan 12;373(6510):109. doi: 10.1038/373109a0. No abstract available. PMID 7816089
- [Background] Ozan E, Okur H, Eker C, Eker OD, Gonul AS, Akarsu N. The effect of depression, BDNF gene val66met polymorphism and gender on serum BDNF levels. Brain Res Bull. 2010 Jan 15;81(1):61-5. doi: 10.1016/j.brainresbull.2009.06.022. PMID 19589373
- [Background] Phillips BE, Kelly BM, Lilja M, Ponce-Gonzalez JG, Brogan RJ, Morris DL, Gustafsson T, Kraus WE, Atherton PJ, Vollaard NBJ, Rooyackers O, Timmons JA. A Practical and Time-Efficient High-Intensity Interval Training Program Modifies Cardio-Metabolic Risk Factors in Adults with Risk Factors for Type II Diabetes. Front Endocrinol (Lausanne). 2017 Sep 8;8:229. doi: 10.3389/fendo.2017.00229. eCollection 2017. PMID 28943861
- [Background] Rovio S, Kareholt I, Helkala EL, Viitanen M, Winblad B, Tuomilehto J, Soininen H, Nissinen A, Kivipelto M. Leisure-time physical activity at midlife and the risk of dementia and Alzheimer's disease. Lancet Neurol. 2005 Nov;4(11):705-11. doi: 10.1016/S1474-4422(05)70198-8. PMID 16239176
- [Background] Schinder AF, Poo M. The neurotrophin hypothesis for synaptic plasticity. Trends Neurosci. 2000 Dec;23(12):639-45. doi: 10.1016/s0166-2236(00)01672-6. PMID 11137155
- [Background] Teri L, Gibbons LE, McCurry SM, Logsdon RG, Buchner DM, Barlow WE, Kukull WA, LaCroix AZ, McCormick W, Larson EB. Exercise plus behavioral management in patients with Alzheimer disease: a randomized controlled trial. JAMA. 2003 Oct 15;290(15):2015-22. doi: 10.1001/jama.290.15.2015. PMID 14559955
- [Background] Vaynman S, Ying Z, Gomez-Pinilla F. Hippocampal BDNF mediates the efficacy of exercise on synaptic plasticity and cognition. Eur J Neurosci. 2004 Nov;20(10):2580-90. doi: 10.1111/j.1460-9568.2004.03720.x. PMID 15548201
- [Background] Unsworth N, Heitz RP, Schrock JC, Engle RW. An automated version of the operation span task. Behav Res Methods. 2005 Aug;37(3):498-505. doi: 10.3758/bf03192720. PMID 16405146
- [Background] Weuve J, Kang JH, Manson JE, Breteler MM, Ware JH, Grodstein F. Physical activity, including walking, and cognitive function in older women. JAMA. 2004 Sep 22;292(12):1454-61. doi: 10.1001/jama.292.12.1454. PMID 15383516